CLINICAL TRIAL: NCT06088992
Title: An Investigator-Initiated Open-Label, Multiple-Dose Clinical Study to Evaluate the Safety,Tolerability, and Efficacy of Gene Therapy for 2Leber's Congenital Amaurosis with RPE65 Mutation (LCA2)
Brief Title: Leber Congenital Amaurosis Inherited Blindness of Gene Therapy Trial(LIGHT)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: HuidaGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Peiquan Zhao, Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG00401; NCT06064565 (obsolete NCT alias)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Leber Congenital Amaurosis
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG004 (Experimental)
  Interventions: Genetic: HG004

INTERVENTIONS:
Genetic: HG004 — Method of Administration: Once unilateralsubretinal injection; The duration of the study isabout 60 weeks for each subject including a 8-weekscreening period, enrollment/baseline visit,treatment visit, and 52 weeks follow-up period.

SUMMARY:
The purpose of the study is to determine whether HG004 as gene therapy is safe and effective for the treatment of Leber Congenital Amaurosis caused by mutationsin RPE65 gene.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between 8 and 50 years of age at the time of signing theinformed consent form.
* Willing to adhere to protocol as evidenced by written informed consent orparental permission and subject assent.
* Clinical confirmed diagnosis of Leber congenital amaurosis (LCA) andmolecular diagnosis of LCA due to RPE65 mutations.
* Ability to perform tests of visual and retinal function.
* Visual acuity of ≤ 20/160 or visual field less than 20 degrees in the eye to beinjected.
* Acceptable hematology, clinical chemistry, and urine laboratory parameters.

Exclusion Criteria:

* OCT examination determined that the outer nuclear layer was not visible inthe planned injection area (Bleb) in the study eye.
* Presence of epiretinal membrane by OCT.
* Complicating systemic diseases or clinically significant abnormal baselinelaboratory values.
* Complicating systemic diseases would include those in which the diseaseitself, or the treatment for the disease, can alter ocular function.
* Prior ocular surgery within six months.
* Prior gene therapy or oligonucleotide therapy treatments.
* Any other condition that would not allow the potential subject to completefollow-up examinations during the study and would, in the opinion of theinvestigator, make the potential subject unsuitable for the study.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and systemic adverse events | 26 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

CONTACTS AND LOCATIONS:
Overall Officials: Peiquan Zhao, Principal Investigator — Xinhua Hospital affiliated with Shanghai Jiao Tong UniversitySchool of Medicine
Locations (1):
- Xinhua Hospital affiliated with Shanghai Jiao Tong UniversitySchool of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No